CLINICAL TRIAL: NCT02147600
Title: Therapeutic Drug Monitoring of Adalimumab in Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC UZG 2013/1148
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis
Keywords: adalimumab; biologicals; immunogenicity
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic plaque psoriasis: Patients suffering from chronic plaque psoriasis, treated with adalimumab (40mg) subcutaneously every other week after an initial dose of 80 mg. Treatment duration of at least 24 weeks.

SUMMARY:
The main goal of this study is to determine optimal cut-off values of adalimumab trough levels corresponding to good clinical response. Determination of these values is necessary to compose a therapeutic algorithm, in which the dosing schedule can be adjusted according to serum trough levels of adalimumab and AAA (anti-adalimumab antibodies). A secondary objective of this study is to further detect and quantify AAA and to correlate them with adalimumab and clinical response in a real life setting cohort of psoriatic patients.

DETAILED DESCRIPTION:
In a multicenter cross-sectional study, 73 adult patients treated with adalimumab (40 mg) every other week for at least 24 weeks are assessed for psoriasis disease severity through measurement of the Psoriasis Area and Severity Index (PASI) before adalimumab treatment start, and prior to sampling. Patients who interrupted their treatment schedule during the 24 weeks prior to blood sampling are excluded. Samples of patients who were treated with adalimumab for any other inflammatory disease and later developed psoriasis are also excluded. Percentage of PASI improvement compared to baseline (∆PASI) represents clinical response. Patients are classified as nonresponders (∆PASI<50), moderate responders (∆PASI 50-75) or good responders (∆PASI 75-100).Serum is collected for adalimumab trough level and anti-drug antibody determination (Sanquin, The Netherlands). By receiver-operator characteristics (ROC) analysis, a cut-off value of adalimumab trough level can be determined to distinguish insufficient from adequate responders.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18 years old
* chronic plaque psoriasis
* adalimumab (40mg) subcutaneously every other week
* at least 24 weeks of adalimumab treatment

Exclusion Criteria:

* interruption of treatment schedule during 24 weeks prior to sampling
* adalimumab for other inflammatory disease and later developed psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Primary care clinic
  * University Hospital
  * Private dermatology practice
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2014-04-10 (Actual); Study Completion 2014-04-10 (Actual)

PRIMARY OUTCOMES:
75% improvement in clinical response | at least 24 weeks of treatment duration
  Minimum of 75 % PASI improvement compared to baseline (∆PASI 75) represents 75% improvement in clinical response.

SECONDARY OUTCOMES:
anti-adalimumab antibody formation | at least 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof.Dr., Study Director — Ghent University, Dpt. of Dermatology; Emma Coussens, Principal Investigator — Ghent University, Dpt. of Dermatology
Locations (5):
- Belgium (5):
  - Ghent University, Dpt. of Dermatology, Ghent
  - Maria Middelares Hospital, Ghent
  - St. Lucas Hospital, Ghent
  - H Hart Hospital, Mol
  - ST Rembert Hospital, Torhout